CLINICAL TRIAL: NCT05038891
Title: Self-Obtained Transperineal and Transvaginal Ultrasound Scans for Measurement of Cervical Dilation and Effacement in Labor: Implications for Telemedicine and Home Hospital in Obstetrics
Brief Title: Self-Obtained Ultrasound Scans for Measurement of Cervical Dilation and Effacement in Labor
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Regan N. Theiler, Associate Professor of Obstetrics and Gynecology, Mayo Clinic
Other Study IDs: 21-004735
Record Dates: First submitted 2021-08-25; First posted 2021-09-09 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Cervical Dilation
Keywords: Cervical Effacement; Cervical Dilation; Labor; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Digital Cervical Assessment performed first: A digital cervical exam will be performed by an experienced senior obstetrics and gynecology resident, using index finger and middle finger to measure the dilation and thickness of the cervix. This is the gold standard measurement utilized to assess the labor course. In this group, the digital cervical exam is done first, followed by a participant-performed ultrasound imaging assessment of the cervix.
  Interventions: Diagnostic Test: Digital Cervical Exam; Diagnostic Test: Transperineal Ultrasound; Diagnostic Test: Transvaginal Ultrasound
- Ultrasound Assessment performed first: Ultrasound imaging will be first taught by an experienced RN, then self-performed by the participant in the presence of junior obstetrics and gynecology resident and the RN. The junior resident will ensure the ultrasound device is functioning properly and the images are saved. In this group, the participant-performed imaging assessment is done first, followed by a digital cervical exam performed by an experienced senior obstetrics and gynecology resident.
  Interventions: Diagnostic Test: Digital Cervical Exam; Diagnostic Test: Transperineal Ultrasound; Diagnostic Test: Transvaginal Ultrasound

INTERVENTIONS:
Diagnostic Test: Digital Cervical Exam — Standard Digital Cervical Exam by an experienced OB provider
Diagnostic Test: Transperineal Ultrasound — Self-administered transperineal ultrasound after instruction by a health care professional
Diagnostic Test: Transvaginal Ultrasound — Self-administered transvaginal ultrasound after instruction by a health care professional

SUMMARY:
This is a pilot study to test the accuracy and comfort of self-directed ultrasound imaging of cervical dilation and effacement in pregnant women undergoing induction of labor. The study will assess correlation of cervical measurements between self-directed imaging and experienced provider digital cervical examinations.

DETAILED DESCRIPTION:
The primary objective will assess correlation of cervical measurements with gold standard of provider digital cervical examinations and self-obtained transperineal and transvaginal images. Experienced providers performing digital cervical examinations will be blinded to ultrasound images and measurements. The maternal-fetal medicine subspecialist interpreting the ultrasound images will be blinded to patient details and will document ultrasound measurement of cervical dilation of the internal cervical os as the mean of anterior-posterior and transverse measurements and cervical length. 2-D ultrasound images and cine clips will be obtained at up to five different time points during the induction of labor.

As as secondary objective, participant discomfort and anxiety will be measured following the initial set of cervical measurements using the Visual Analog Scale and Six-Item State-Trait Anxiety Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females age 18 years or older
* Third trimester of pregnancy with a singleton fetus (gestational age >28 weeks)
* Pre-gestational body mass index <40
* Scheduled for induction of labor
* Eligible for induction of labor based on current birth center guidelines
* Intact membranes when presenting for induction of labor

Exclusion Criteria:

* History of prior cervical loop electrosurgical excisional procedure or cold knife conization
* Cerclage placement during current pregnancy
* Positive COVID-19 test within 7 days of admission for induction of labor
* Fever > 38.0 C at time of admission for induction of labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This pilot study will enroll pregnant women undergoing induction of labor at the Family Birth Center at Mayo Clinic Hospital in Rochester, MN. The target population will include women with a singleton fetus at gestational age greater than 28 weeks 0 days gestation who have intact membrane status at time of induction of labor.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Correlation of cervical examination between self-obtained ultrasound measurements and provider digital exam. | Data collection during induction of labor with image interpretation through end of study, assessed up to 6 months
  Data collection will occur at up to five time points along a participant's labor course. Providers will be blinded to ultrasound images. Data includes provider digital exam, transperineal ultrasound cine clip with mean (anterior-posterior and transverse) measurement of internal os and total cervical length and transvaginal ultrasound cine clips with mean (anterior-posterior and transverse) measurement of internal os and total cervical length. Ultrasound images will be read by maternal-fetal medicine subspecialist blinded to patient information, labor stage and provider cervical examination.

SECONDARY OUTCOMES:
Participant-perceived discomfort after cervical examination using a 10 point Visual Analog Scale (VAS) | On day of induction after first cervical examination during first assessment, through study completion up to 6 months
  The Visual Analog Scale values range from 0 to 10 where higher values indicate more pain and will be assessed once after the first cervical examination.
Participant anxiety levels will be measured via the Six-Item Spielberger State-Trait Anxiety Inventory (STAI-6) | On day of induction after first cervical examination during first assessment, through study completion up to 6 months
  The 6 items which are on a 4 point likert scale will be administered to participants post first cervical exam. The 6 items are summed, divided by 6 and hen multiplied by 20 to give a range of 20 to 80. Higher scores indicate more anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Regan N Theiler, M.D., Principal Investigator — Mayo Clinic; Megan Miller, M.D., Study Chair — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Mayo Clinic Methodist Hospital, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials